CLINICAL TRIAL: NCT03805893
Title: Investigation of Plastic Changes in the CNS Associated With Peripheral Neuropathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Otto Muzik, Professor of Pediatrics, Wayne State University
Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1811001903
Record Dates: First submitted 2019-01-08; First posted 2019-01-16 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Peripheral Neuropathy
MeSH Terms: conditions — Peripheral Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: Two groups: patients with peripheral neuropathy and normal controls
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Moderate heat pain — To apply a sensory challenge that can be applied over longer periods required for PET imaging and that is also compatible with high magnetic fields during MRI scanning, we will use a well-established thermal challenge of the lower extremity. To apply mildly painful heat to the patient, the right leg (from the foot up to the knee) will be wrapped in a blanket that incorporates a network of small-diameter plastic tubing through which hot water (45 - 55 oC) is circulated from a temperature-controlled reservoir.

SUMMARY:
Recent neuroimaging literature on neuropathy suggests that chronic pain is characterized by learning-related and memory-related plastic changes of the central nervous system (CNS) with concomitant maladaptive changes in body perception. In particular, it is well accepted that learning-induced functional and structural brain changes involve, in addition to sensorimotor cortex, also limbic and frontal areas that mediate the transition from acute to chronic pain, resulting in pathological processing of body image, impaired multisensory integration and faulty feedback from various interoceptive processes. Interestingly, these alterations share many similarities with brain changes in emotional disorders and the specificity for pain needs to be determined. Moreover, the diagnosis and management of neuropathic pain syndromes remains a major clinical challenge, and this failure is partly attributed to our inability to identify functional brain changes that not only contribute to these syndromes, but also expose the patient to psychological burden that might lead to drug abuse. Although opioids are currently used frequently as first line therapy to alleviate pain caused by the various forms of neuropathies, recent reports indicate that long-term opioid therapy does not improve functional status but rather is associated with a higher risk of depression as well as subsequent opioid dependency and overdose. Thus, in order to improve therapeutic interventions in this patient group, it is imperative to develop a mechanistic model of central processes that could both explain and predict longitudinal changes associated with neuropathic pain syndromes. The identification of the correct sources of pain sensation (i.e. the contribution of central rather than peripheral factors to pain chronicity) is of paramount importance since the clinical course and patient management is likely to differ depending on the exact underlying cause.

DETAILED DESCRIPTION:
The goal is to relate non-invasive brain imaging data to clinical parameters in order to develop a mechanistic model of CNS adaptive processes that are produced by a patient-specific disease state. The investigators believe that such a model will have significant predictive value and might provide added value for subsequent patient management. To achieve the stated objectives, the following Specific Aim will be tested:

Aim 1. To assess regional brain changes in patients with polyneuropathies associated with a mild thermal pain challenge and to relate these changes to clinical measures of neuropathy.

Hypothesis 1A. Regional changes in brain glucose metabolism (as measured using FDG PET/CT imaging) associated with thermal pain will differ between patients with polyneuropathy and a group of age-matched controls. Specifically, patients with neuropathy will show a significantly higher increase in glucose metabolism in the medial pain system (affective dimension - brainstem, amygdala, insula) following thermal pain as compared to the control group, indicating increased sensitivity of the interoceptive neural control system for peripheral pain stimulation in patients.

Hypothesis 1B. In patients with neuropathy, regional changes in brain glucose metabolism associated with thermal pain in the medial pain system (affective dimension - brainstem, amygdala, insula) will be inversely related to clinical measures of neuropathic disease state (as measured using quantitative sensory testing, nerve conduction study and standardized pain scale assessment). In contrast, glucose metabolic changes in the lateral pain system (discriminatory dimension - thalamus, area S1) will be directly related to clinical measures. The extent of changes in the medial versus lateral system will also be correlated with the types of polyneuropathies, including idiopathic painful sensory neuropathy, chronic inflammatory demyelinating polyneuropathy (CIDP) and Charcot-Marie-Tooth type-1A (CMT1A, the most common type of inherited peripheral nerve disease).

Hypothesis 1C. The increase in functional connectivity (as assessed using fMRI following an oscillatory thermal pain paradigm) will differ between neuropathic patients and controls. Specifically, functional connectivity between the medial pain system (brainstem, amygdala, insula) and the cognitive pain system (VLPFC and FP) will be significantly higher in the patient group as compared to the controls, indicating increased inhibition of the interoceptive brain network by the executive control system. Moreover, functional connectivity between the medial and cognitive pain systems will be directly related with clinical measures.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of a peripheral nerve disease - IPN, CIDP or CMT1A (patient group only)
2. Healthy volunteers with no history of medical conditions known to afflict the nervous system will be recruited as normal controls (control group only)
3. Age 18-60 (Inclusive)
4. Able to undergo PET and MRI
5. Patients who are not on sedative, antidepressant, sedative antihistaminic or narcotic medications.

Exclusion Criteria:

1. Any subject unwilling to undergo genetic testing (DNA sampling)
2. Any subjects with history of conditions known to affect the PNS, such as diabetes, stroke, thyroid disease, chemotherapy, renal failure, alcohol abuse, etc.
3. Subjects with abnormal physical findings suggesting peripheral nerve diseases.
4. Subjects of reproductive potential, who are sexually active but unwilling and/or unable to use medically appropriate contraception, or women who are pregnant or breastfeeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-02-01 (Estimated); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Regional brain glucose metabolic changes | Day 0
  Changes in brain glucose metabolism associated with thermal pain in the brainstem, amygdala and insula regions. Units are the % change in regional standard uptake value (SUV) between the control and the thermal pain PET scan.
Nerve conduction assessment | Day 0
  Electromyography (EMG) study determining nerve conduction velocity (NCV). The unit of NCV is m/s. The lower the NCV values, the more severe is the neuropathy.
Pain Scale Assessment | Day 0
  Neuropathy Pain Scale (NPS) instrument. Units is a score between 0 (no pain) and 100 (worst possible pain).

IPD SHARING:
Plan to Share IPD: No
Results of the study will be published in international journals.